CLINICAL TRIAL: NCT03704103
Title: mHealth Insulin Titration and Management (iSage)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00142758
Record Dates: First submitted 2018-08-28; First posted 2018-10-12 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iSage for adjustment of insulin (Experimental): The provider will prescribe the iSage app to the subject and choose a treatment algorithm within the app to make insulin dose adjustments.
  Interventions: Other: iSage
- Conventional management (No Intervention): Our clinic uses a modified treat-to-target algorithm which is summarized on a 3 x 5 refrigerator magnet.

INTERVENTIONS:
Other: iSage — The provider will choose a treatment algorithm within the iSage app and set the parameters to make insulin dose adjustments no less frequently than every 7 days. The patient is instructed to perform daily fasting glucose measurements and follow the app's recommendations for insulin adjustment.
  Arms: iSage for adjustment of insulin

SUMMARY:
The purpose of this study is to determine the benefits of using the iSage app for basal insulin titration and support. By doing this study the investigators hope to learn whether the app improves the participant's ability to follow his/her healthcare provider's instructions to adjust his/her insulin doses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Type 2 Diabetes, based on the World Health Organization (WHO) criteria, treated with basal insulin
* HbA1c 8-11% inclusive
* Glomerular filtration rate (GFR) > 60 ml/min
* Has an Android or iOS based compatible smartphone (iOS 9.0 or above, Android 4.4 or above)
* Willing to perform at least 1 fasting finger stick glucose measurements every morning
* English speaking

Exclusion Criteria:

* Diagnosis of hypoglycemic unawareness
* Diagnosis of hyperglycemic hyperosmolar non-ketotic coma (HONK) or diabetic ketoacidosis (DKA) within 6 months of enrollment
* Recent (within the last 6 months)/current use of non-topical steroids
* Insulin requirements in excess of 1 U/kg per day
* Use of pioglitazone or another thiazolidinedione (TZD)
* In the opinion of the provider, HgbA1c goals should be adjusted above 7% due to infirmity, unstable cardiovascular disease, etc.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Concentration of HgbA1c | 90 days
  The investigators will compare changes in HgbA1c from baseline to day 90.
Number of participants meeting HgbA1c <7% | 90 days
  The investigators will calculate the percent of patients achieving HgbA1c <7% at day 90.

SECONDARY OUTCOMES:
Sustained use of the iSage app (iSage group only) | 90 days
  The investigators will compare the percentage of subjects using the app as prescribed versus "dropouts".
Hypoglycemia | 90 days
  The investigators will record the number of episodes of hypoglycemia, to include severity of event, related symptoms, and time of day.

OTHER OUTCOMES:
Healthcare resource utilization | 90 days
  Number of contacts with healthcare resources (including telephone calls), ER visits, clinic visits, hospitalizations
Diabetes Quality of Life Survey (DQOL) | 90 days
  The investigators will compare DQOL scores from baseline to day 90. The 15-item DQOL Brief Clinical Inventory provides a total health-related quality of life score that predicts self-reported diabetes care behaviors and satisfaction with diabetes control as effectively as the full version of the instrument. Items are scored on a 5-point Likert scale and are of two general formats. One format asks about the frequency of negative impact of diabetes itself or of the diabetes treatment (i.e., "How often do you worry about whether you will pass out?") and provides response options from 1 (never) to 5 (all the time). The second format asks about satisfaction with treatment and quality of life (i.e., "How satisfied are you with the time you spend exercising?") and is scored from 1 (very satisfied) to 5 (very dissatisfied). Higher scores are negatively valanced, indicating problem frequency or dissatisfaction.
Insulin Treatment Satisfaction Questionnaire (ITSQ) | 90 days
  The investigators will compare ITSQ scores from baseline to day 90. The 22-item ITSQ is applicable to a wide variety of insulin therapies, and measures insulin treatment satisfaction assessing regimen inconvenience, lifestyle flexibility, glycemic control, hypoglycemic control, and satisfaction with the insulin delivery device. The response scale is ordinal, ranging from 1 (extremely satisfied) to 6 (extremely dissatisfied). The ITSQ is scored among 5 content clusters, forming a total ITSQ score between 0% to 100%, where 100% indicates complete satisfaction with insulin treatment.
iSage Product Satisfaction Survey (iSage group only) | 90 days
  The investigators will assess iSage app ease of use and satisfaction. Survey consists of 3 items. Answer choices range from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States